CLINICAL TRIAL: NCT04959955
Title: Project to Improve the Diagnosis and Treatment Ability of Adult Severe Community Acquired Lower Respiratory Tract Infection
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: First Hospital of China Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: LM2016057
Record Dates: First submitted 2021-07-04; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: CAP; COPD Exacerbation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AECOPD group
- CAP group

INTERVENTIONS:
Diagnostic Test:

SUMMARY:
1. Objective to understand the proportion of atypical pathogens in the pathogens of SCAP and AECOPD in urban hospitals in China.
2. Objective to investigate the antimicrobial resistance of atypical pathogens in patients with acute exacerbation of chronic obstructive pulmonary disease (COPD) and SCAP in urban hospitals.
3. Objective to master the important clinical characteristics of patients with acute exacerbation of SCAP and COPD caused by atypical pathogens and mixed infection in urban hospitals in China, and to put forward the experience judgment index.
4. Objective to evaluate the advantages of various diagnostic methods for atypical pathogens causing lower respiratory tract infection.
5. It is suggested that the current empirical treatment of SCAP and severe COPD in China should be improved.

ELIGIBILITY:
Inclusion Criteria:

* SCAP
* AECOPD

Exclusion Criteria:

* Pregnant or lactating women.

  * Patients with bronchiectasis.

    * Patients with active pulmonary tuberculosis.

      * Aspiration pneumonia or obstructive pneumonia.

        * Two weeks before the onset of hospital treatment history, this infection can not be excluded from hospital acquired infection.

          * HIV positive patients (but HIV testing is not required).

            * Patients who are unable and / or unable to understand and / or implement the investigation protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult hospitalized cases of SCAP and acute exacerbation of COPD were collected from 12 medical institutions in 10 cities in China within 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-08-08 (Actual); Primary Completion 2016-07-10 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Incidence of atypical pathogens and mixed infections | 2year Incidence
  Incidence of atypical pathogens and mixed infections

IPD SHARING:
Plan to Share IPD: No